CLINICAL TRIAL: NCT06899061
Title: A Modular Phase I, Open-label Study to Assess the Safety, Pharmacokinetics, and Drug Interaction Potential and Relative Bioavailability of Saruparib in Patients With Advanced Solid Malignancies
Brief Title: Modular Clinical Pharmacology Study to Evaluate the Drug-drug Interaction Potential and Relative Bioavailability of Saruparib
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D9723C00002; 2024-513692-41-00 (Registry Identifier: EUCTR)
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Malignancies
Keywords: Single-stranded DNA; Poly(ADP-ribose) polymerase 1; Transporter substrates; Pharmacokinetics
MeSH Terms: interventions — Digoxin; ATP Binding Cassette Transporter, Subfamily B, Member 1; Furosemide; Metformin; Rosuvastatin Calcium; Rabeprazole

STUDY DESIGN:
Intervention Model Description: Module 1: Single Group Module 2: Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Cohort (Module 1) (Active Comparator): Period 1: participants will receive a single oral dose of cocktail substrate (digoxin, furosemide, metformin hydrochloride, and rosuvastatin) on Day 1.
  Period 2: participants will receive a single dose saruparib from Day 1 to 9, and a single dose of cocktail substrate on Day 5 in combination with saruparib.
  Period 3: participants will receive a single oral dose of saruparib daily.
  Interventions: Drug: Saruparib; Drug: Digoxin; Drug: Furosemide; Drug: Metformin Hydrochloride; Drug: Rosuvastatin
- Saruparib RC Cohort (Module 2) (Active Comparator): Period 1: participants will receive a single dose of RC saruparib. Period 2: participants will receive a single dose of DC saruparib. Period 3: participants will receive rabeprazole twice daily from Day 1 to 3, and a single dose of rabeprazole prior to DC saruparib on Day 4.
  Period 4: participants will receive RC saruparib daily for up to 3 cycles.
  Interventions: Drug: Saruparib; Drug: Rabeprazole
- Saruparib DC Cohort (Module 2) (Active Comparator): Period 1: participants will receive a single dose of DC saruparib. Period 2: participants will receive a single dose of RC saruparib. Period 3: participants will receive rabeprazole twice daily from Day 1 to 3, and a single dose of rabeprazole prior to DC saruparib on Day 4.
  Period 4: participants will receive RC saruparib daily for up to 3 cycles.
  Interventions: Drug: Saruparib; Drug: Rabeprazole

INTERVENTIONS:
Drug: Saruparib — Module 1:
  Period 2: participants will receive saruparib orally once daily from Day 1 to Day 9. On Day 5 saruparib will be administered orally in combination with the cocktail of substrates.
  Period 3: participants will receive saruparib orally once daily for up to 3 cycles of 28 days each.
  Module 2:
  Period 1 and Period 2: participants will receive a single oral dose of DC or RC saruparib.
  Period 3: participants will receive an oral dose of rabeprazole twice daily from Day 1 to 3, and a single oral dose of rabeprazole prior to DC saruparib on Day 4.
  Period 4: participants will receive an oral dose of RC saruparib daily for 3 cycles.
Drug: Digoxin — Period 1: participants will receive a single oral dose of a cocktail of substrates (digoxin, furosemide, metformin hydrochloride, and rosuvastatin) on Day 1.
  Period 2: participants will receive a single oral dose of the cocktail of substrates in combination with saruparib on Day 5.
  Other Names: P-gp
  Arms: Treatment Cohort (Module 1)
Drug: Furosemide — Period 1: participants will receive a single oral dose of a cocktail of substrates (digoxin, furosemide, metformin hydrochloride, and rosuvastatin) on Day 1.
  Period 2: participants will receive a single oral dose of the cocktail of substrates in combination with saruparib on Day 5.
  Other Names: OCT2
  Arms: Treatment Cohort (Module 1)
Drug: Metformin Hydrochloride — Period 1: participants will receive a single oral dose of a cocktail of substrates (digoxin, furosemide, metformin hydrochloride, and rosuvastatin) on Day 1.
  Period 2: participants will receive a single oral dose of the cocktail of substrates in combination with saruparib on Day 5.
  Other Names: OAT1/3, MATE1/2K
  Arms: Treatment Cohort (Module 1)
Drug: Rosuvastatin — Period 1: participants will receive a single oral dose of a cocktail of substrates (digoxin, furosemide, metformin hydrochloride, and rosuvastatin) on Day 1.
  Period 2: participants will receive a single oral dose of the cocktail of substrates in combination with saruparib on Day 5.
  Other Names: OATP1B1/3
  Arms: Treatment Cohort (Module 1)
Drug: Rabeprazole — Period 3: Participants will receive two doses of rabeprazole per day from Day 1 to 3. On Day 4, participants will receive a dose of rabeprazole followed by DC saruparib.
  Arms: Saruparib DC Cohort (Module 2); Saruparib RC Cohort (Module 2)

SUMMARY:
A Phase I modular study to assess the effect of oral saruparib on other treatments in patients with advanced solid malignancies.

DETAILED DESCRIPTION:
Module 1 of the study is a Phase I, open-label study to assess the effects of saruparib on the PK of substrates digoxin (P-gp), furosemide (OAT1/3), metformin hydrochloride (OCT2/MATE1/2K), and rosuvastatin (OATP1B1/3) in participants with advanced solid malignancies.

Module 2 of the study is a Phase I, open-label, 4-treatment period, multi-centre, relative bioavailability, PPI effect, randomised, crossover study of saruparib tablets manufactured using a direct compression (DC) process in participants with advanced solid malignancies.

Module 1 of the study will include:

* A Screening period of 28 days prior to Day 1.
* Period 1: a single dose of a cocktail of substrates (digoxin, furosemide, metformin hydrochloride, and rosuvastatin) on Day 1.
* A washout period of 1 to 3 days between Period 1 and Period 2.
* Period 2: continuous dosing of saruparib from Day 1 to Day 9. On Day 5 saruparib will be administered in combination with the cocktail of substrates.
* Period 3: a dose of saruparib per day for up to 3 cycles of 28 days each.
* An End of Study visit up to 3 days after the last dose in Period 3.

Module 2 of the study will include:

* A Screening period of 28 days prior to Day 1.
* Period 1 and Period 2: a single dose of roller compaction (RC) or DC saruparib.
* Period 3: from Day 1 to 3, two doses of rabeprazole per day. On Day 4, a dose of rabeprazole followed by DC saruparib.
* A washout period of at least 3 days between Period 1 and Period 3, and between Period 2 and Period 3.
* Period 4: a single dose of RC saruparib for up to 3 cycles.
* An End of Study visit up to 3 days after the last dose in Period 4.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with documented evidence of locally advanced unresectable or metastatic solid tumours, excluding lymphoma, who have exhausted standard of care options (or for which no standard therapies exist) and may be suitable for saruparib monotherapy treatment in the opinion of the investigator.
2. Adequate organ and marrow function (in the absence of transfusions or growth factor support within 28 days prior to enrolment).
3. An ECOG PS: 0 to 1 with no deterioration within 1 week prior to the screening visit.
4. Life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. Evidence of active and uncontrolled hepatitis B and/or hepatitis C. Screening for hepatitis B and hepatitis C is not required, criteria is based on medical history.
2. Participants with controlled HIV need to meet the following criteria (screening for HIV is not required, criteria are based on medical history):

   1. Undetectable viral RNA load less than 400 copies/mL in the last 4 weeks prior to first dose of study intervention.
   2. CD4+ count of ≥ 350 cells/μL.
   3. No history of acquired immunodeficiency syndrome-defining opportunistic infection within the past 12 months, and stable on the same anti-HIV medications for at least 6 months. Screening for HIV is not required.
3. Any other evidence of diseases, such as severe or uncontrolled systemic diseases or active uncontrolled infections, including but not limited to uncontrolled major seizure disorder, active bleeding diseases, superior vena cava syndrome, or history of allogenic organ transplant
4. Active tuberculosis infection
5. Any of the following cardiac criteria:

   1. Mean resting QTcF > 470 ms obtained from triplicate ECGs performed at screening and averaged. At each timepoint at which triplicate ECG are required, 3 individual ECG tracings should be obtained in succession, no more than 2 minutes apart. The full set of triplicates should be completed within 5 minutes.
   2. Any factors that increase the risk of QT prolongation, shortening or risk of arrhythmic events such as hypokalaemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in an immediate family member.
6. History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted if deemed medically safe by the investigator.
7. Other cardiovascular diseases with the exception of alopecia, and peripheral neuropathy; any unresolved toxicities from prior anticancer therapy greater than CTCAE Grade 1 at the time of study enrolment.
8. Any known history of persisting (> 2 weeks) severe pancytopenia due to any cause (absolute neutrophil count < 0.5 × 109/L or platelets < 50 × 109/L).
9. Spinal cord compression, or brain metastases for at least 4 weeks prior to start of study intervention unless asymptomatic and stable (ie, not requiring a dose of steroids ≥ 10 mg for more than 2 weeks). A minimum of 2 weeks must have elapsed between the end of brain radiotherapy and signing the main study ICF.
10. Participants with any known predisposition to bleeding (eg, active peptic ulceration, recent [within 6 months] haemorrhagic stroke, proliferative diabetic retinopathy).
11. Participants with history of MDS/AML or with features suggestive of MDS/AML (as determined by prior diagnostic investigation). If there is no clinical MDS/AML suspicion, no specific screening for MDS/AML is required.
12. Refractory nausea and vomiting, chronic GI diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of study intervention.
13. Known allergy or hypersensitivity to study intervention or any of the excipients of the study intervention.
14. Any condition that, in the opinion of the investigator, would interfere with evaluation of the study intervention or interpretation of participant safety or study results.
15. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
16. Uncontrolled intercurrent illness within the last 12 months, including but not limited to, serious chronic GI conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the participant to give written informed consent.

Module 1:

1. Current or planned use of calcium channel blockers up to the end of Period 2.
2. Current and/or regular use of any of the study interventions in the cocktail substrates that cannot be substituted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
Module 1: Area under plasma concentration-time curve from zero extrapolated to infinity (AUCinf) of digoxin, furosemide, metformin and rosuvastatin when dosed alone and in combination with saruparib | Period 1: Days 1 to 5. Period 2: Days 5 to 9
  To evaluate the effects of saruparib on the PK of substrates of human drug transporters digoxin, furosemide, metformin hydrochloride, and rosuvastatin in participants with advanced solid malignancies.
Module 1: Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) of digoxin, furosemide, metformin and rosuvastatin when dosed alone and in combination with saruparib | Period 1: Days 1 to 5. Period 2: Days 5 to 9
  To evaluate the effects of saruparib on the PK of substrates of human drug transporters digoxin, furosemide, metformin hydrochloride, and rosuvastatin in participants with advanced solid malignancies.
Module 1: Maximum observed plasma (peak) drug concentration (Cmax) of digoxin, furosemide, metformin and rosuvastatin when dosed alone and in combination with saruparib | Period 1: Days 1 to 5. Period 2: Days 5 to 9
  To evaluate the effects of saruparib on the PK of substrates of human drug transporters digoxin, furosemide, metformin hydrochloride, and rosuvastatin in participants with advanced solid malignancies.
Module 2: AUClast between DC and RC tablets of saruparib | Period 1: Days 1 to 3. Period 2: Days 1 to 3
  To assess the relative bioavailability of saruparib tablets manufactured using a DC process versus RC process under fasted conditions.
Module 2: AUCinf between DC and RC tablets of saruparib | Period 1: Days 1 to 3. Period 2: Days 1 to 3
  To assess the relative bioavailability of saruparib tablets manufactured using a DC process versus RC process under fasted conditions.
Module 2: Cmax between DC and RC tablets of saruparib | Period 1: Days 1 to 3. Period 2: Days 1 to 3
  To assess the relative bioavailability of saruparib tablets manufactured using a DC process versus RC process under fasted conditions.
Module 2: AUClast of DC saruparib tablets in the presence and absence of rabeprazole relative to the RC tablet | Period 3: Days 4 to 6
  To evaluate the effect of rabeprazole on saruparib PK profile following the administration of saruparib DC tablets.
Module 2: AUCinf of DC saruparib tablets in the presence and absence of rabeprazole relative to the RC tablet | Period 3: Days 4 to 6
  To evaluate the effect of rabeprazole on saruparib PK profile following the administration of saruparib DC tablets.
Module 2: Cmax of DC saruparib tablets in the presence and absence of rabeprazole relative to the RC tablet | Period 3: Days 4 to 6
  To evaluate the effect of rabeprazole on saruparib PK profile following the administration of saruparib DC tablets.

SECONDARY OUTCOMES:
Module 1: Time to reach peak or maximum observed concentration following drug administration (tmax) of digoxin, furosemide, metformin and rosuvastatin when administered alone and in combination with saruparib, in plasma | Period 1: Days 1 to 5. Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) of digoxin, furosemide, metformin and rosuvastatin when administered alone and in combination with saruparib, in plasma | Period 1: Days 1 to 5. Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of digoxin, furosemide, metformin and rosuvastatin when administered alone and in combination with saruparib, in plasma | Period 1: Days 1 to 5. Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: Volume of distribution (apparent) at steady state following extravascular administration (based on terminal phase) (Vz/F) of digoxin, furosemide, metformin and rosuvastatin when administered alone and in combination with saruparib, in plasma | Period 1: Days 1 to 5. Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: Area under concentration time curve in the dosing interval (AUCtau) of saruparib after multiple doses in plasma | Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: AUClast of saruparib after multiple doses in plasma | Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: Minimum blood plasma concentration reached during a dosing interval (Cmin) of saruparib after multiple doses in plasma | Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Screening (Day -28) to Follow up, up to 129 days
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: Cmax of saruparib after multiple doses in plasma | Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: CL/F of saruparib after multiple doses in plasma | Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: Vz/F of saruparib after multiple doses in plasma | Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: t1/2λz of saruparib after multiple doses in plasma | Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 1: tmax of saruparib after multiple doses in plasma | Period 2: Days 5 to 9
  To assess PK, safety and tolerability of saruparib following oral dosing.
Module 2: Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Screening (Day -28) to Follow up, up to 167 days
  To assess the safety and tolerability of saruparib.
Module 2: Cmax of saruparib via DC and RC tablets | Period 1: Days 1 to 3. Period 2: Days 1 to 3
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: tmax of saruparib via DC and RC tablets | Period 1: Days 1 to 3. Period 2: Days 1 to 3
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: t½λz of saruparib via DC and RC tablets | Period 1: Days 1 to 3. Period 2: Days 1 to 3
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: λz of saruparib via DC and RC tablets | Period 1: Days 1 to 3. Period 2: Days 1 to 3
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: CL/F of saruparib via DC and RC tablets | Period 1: Days 1 to 3. Period 2: Days 1 to 3
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: Vz/F of saruparib via DC and RC tablets | Period 1: Days 1 to 3. Period 2: Days 1 to 3
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: Cmax of saruparib via DC tablets in the presence of rabeprazole | Period 3: Days 4 to 6
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: tmax of saruparib via DC tablets in the presence of rabeprazole | Period 3: Days 4 to 6
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: t½λz of saruparib via DC tablets in the presence of rabeprazole | Period 3: Days 4 to 6
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: λz of saruparib via DC tablets in the presence of rabeprazole | Period 3: Days 4 to 6
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: CL/F of saruparib via DC tablets in the presence of rabeprazole | Period 3: Days 4 to 6
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.
Module 2: Vz/F of saruparib via DC tablets in the presence of rabeprazole | Period 3: Days 4 to 6
  To compare the PK of saruparib manufactured using a DC process versus RC process in participants with advanced solid malignancies.

CONTACTS AND LOCATIONS:
Locations (4):
- Research Site, Sofia, Bulgaria
- Research Site, Chisinau, Moldova
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/